CLINICAL TRIAL: NCT01578525
Title: Medication Safety of Elderly Patients in Hospital and Ambulatory Setting Considering the Transitions of Care for Home-cared Patients and Nursing Home Residents
Brief Title: Medication Safety of Elderly Patients in Hospital and Ambulatory Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Collaborators: Apothekerstiftung Nordrhein, Duesseldorf (Unknown); Foerderinitiative Pharmazeutische Betreuung e.V., Berlin (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11-192
Record Dates: First submitted 2012-04-13; First posted 2012-04-17 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2012-05

CONDITIONS: Elderly; Pharmaceutical Care; Hospital Readmission; Health Services for the Aged; Medication Safety
Keywords: medication safety; elderly; pharmaceutical care; hospital readmission; drug-related readmission; Health Services for the Aged
MeSH Terms: interventions — Pharmaceutical Services

ARMS (2):
- standard care (No Intervention): Standard care (by German definition), traditional care by physician and nurse on the ward
- Intensified standard care (Other): Intensified standard care: traditional care by physician and nurse, additional pharmaceutical care by a pharmacist during hospitalization
  Interventions: Other: Pharmaceutical Care Service

INTERVENTIONS:
Other: Pharmaceutical Care Service — Checking medication under safety considerations (medication at admission, hospitalization, discharge); recommendations for potentially inappropriate medication (PRISCUS-criteria),
  Arms: Intensified standard care

SUMMARY:
The purpose of this study is to determine whether additional pharmaceutical care for elderly patients (home-cared patients, nursing-home residents) has a positive impact on drug-related readmissions.

ELIGIBILITY:
Inclusion Criteria:

* patient 65 years old or older
* patient admitted to one of the project wards
* minimum hospitalization: 3 days
* written informed consent (patient or the legal representative)
* current medication of the patient at hospitalization

Exclusion Criteria:

* patients included in this study previously

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 61 (Actual)
Dates: Start 2012-04; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Drug-related readmission | one year after discharge from the cooperating ward

SECONDARY OUTCOMES:
Adverse drug events | during hospital stay on cooperating wards(continuous data collection during routine ward rounds;hence,duration of data collection is dependent on individual hospital stay of each patient, up to 1 year) and 1 year after discharge from the cooperating ward
Number of prescribed potentially inappropriate medication (PRISCUS-criteria) | during hospital stay on cooperating wards(continuous data collection during routine ward rounds;hence,duration of data collection is dependent on individual hospital stay of each patient, up to 1 year) and 1 year after discharge from the cooperating ward
  The PRISCUS list was developed in 2010 for the German market. Potentially inappropriate medications were judged as inappropriate by an expert panel using the Delphi technique. [Holt et al., Dtsch Arztebl 2010]
time to readmission | one year after discharge from the cooperating ward
Number of accepted recommendations in the intervention group | during hospital stay on cooperating wards (continuous data collection during routine ward rounds; hence, duration of data collection is dependent on individual hospital stay of each patient, up to one year) in the intervention group
time for intervention | during hospital stay on cooperating wards (continuous data collection during routine ward rounds; hence, duration of data collection is dependent on individual hospital stay of each patient, up to one year) in the intervention group
  time recording for pharmaceutical care service
drug-related problem | during hospital stay on cooperating wards (continuous data collection during routine ward rounds; hence, duration of data collection is dependent on individual hospital stay of each patient, up to one year) in the intervention group
number of changes in medication after discharge | one year

CONTACTS AND LOCATIONS:
Overall Officials: Albrecht Eisert, Dr. rer. nat., Study Director — University Hospital Aachen, Hospital Pharmacy, Steinbergweg 20, 52074 Aachen, Germany; Axel Heidenreich, Prof. Dr. med., Principal Investigator — University Hospital Aachen, Department of Urology, Pauwelsstr. 30, 50274 Aachen, Germany; Joerg B Schulz, Prof. Dr. med., Principal Investigator — University Hospital Aachen, Department of Neurology, Pauwelsstr. 30, 52074 Aachen, Germany; Christian Trautwein, Prof. Dr. med., Principal Investigator — University Hospital Aachen, Internal Medicine III (Gastroenterology and Metabolic Disorders), Pauwelsstr. 30, 52074 Aachen, Germany; Ulrich Jaehde, Prof. Dr. rer. nat., Study Chair — University of Bonn, Pharmaceutical Institute, Clinical Pharmacy, An der Immenburg 4, 53121 Bonn, Germany; Rebekka Heumueller, Principal Investigator — University Hospital Aachen, Hospital Pharmacy, Steinbergweg 20, 52074 Aachen, Germany; Nicolaus Marx, Prof. Dr. med., Principal Investigator — University Hospital Aachen,Internal Medicine I (Cardiology, Pneumology, Angiology and Internal Intensive Medicine)
Locations (1):
- University Hospital Aachen, Aachen, Germany

REFERENCES:
- [Derived] Lenssen R, Schmitz K, Griesel C, Heidenreich A, Schulz JB, Trautwein C, Marx N, Fitzner C, Jaehde U, Eisert A. Comprehensive pharmaceutical care to prevent drug-related readmissions of dependent-living elderly patients: a randomized controlled trial. BMC Geriatr. 2018 Jun 4;18(1):135. doi: 10.1186/s12877-018-0814-3. PMID 29898670